CLINICAL TRIAL: NCT00404339
Title: Adjuvant p53 Peptide Loaded DC-Based Therapy for Subjects With Squamous Cell Cancer of the Head and Neck (A Phase I Safety and Immunogenicity Trial)
Brief Title: Vaccine Therapy in Treating Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Ferris (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Robert Ferris, UPMC Endowed Professor and Chief, Division of Head and Neck Surgery, Department of Otolaryngology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCI-03-156; CDR0000515081 (Registry Identifier: PDQ (Physician Data Query)); PCI-0507062; NCT00235612 (obsolete NCT alias)
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: mutant p53 peptide pulsed dendritic cell vaccine
Biological: tetanus toxoid helper peptide
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Vaccines made from a person's dendritic cells mixed with peptides may help the body build an effective immune response to kill tumor cells.

PURPOSE: This randomized phase I trial is studying the side effects of vaccine therapy in treating patients with head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity of intranodally injected autologous dendritic cells (DC) loaded with wild-type p53 peptides with or without T-helper peptide epitope in patients with squamous cell carcinoma of the head and neck.

Secondary

* Determine the local and systemic immunomodulatory effects of this vaccine in these patients.

OUTLINE: This is a randomized, pilot study.

Patients undergo leukapheresis. The resulting dendritic cells (DC) are pulsed with wild-type (wt) p53 peptides with or without T-helper (Th) peptides. Individual autologous vaccines are prepared for each patient. Patients who are HLA-A2-DR4-negative are randomized to 1 of 2 treatment arms (arm I or arm II). Patients who are HLA-A2-DR4-positive are assigned to arm III.

* Arm I: Patients receive autologous DC loaded with HLA-A2.1-restricted wt p53 peptides only.
* Arm II: Patients receive autologous DC loaded with HLA-A2.1-restricted wt p53 peptides and Th tetanus toxoid peptide.
* Arm III (HLA-A2-DR4-positive patients only): Patients receive autologous DC loaded with HLA-A2.1-restricted wt p53 peptides and Th wt p53 peptide.

In all arms, each vaccine is administered by ultrasonography-guided inguinal intranodal injection over 30 minutes on days 0, 14, and 28.

After completion of study therapy, patients are followed periodically.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck

  * Resectable disease
  * Any stage allowed
* Successfully treated with curative intent
* Recurrent disease allowed provided the following criteria are met:

  * No evidence of disease
  * At least 6 weeks since prior antitumor therapy
* Positive for HLA-A2.1

  * HLA-DR4 allele status known
* Tumor tissue must be available
* No active brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0 or 1
* Life expectancy ≥ 6 months
* Granulocyte count > 2,500/mm^3
* Lymphocyte count > 700/mm^3
* Platelet count > 100,000/mm^3
* Bilirubin < 0.2 mg/dL
* Creatinine < 0.2 mg/dL
* Hemoglobin > 8 g/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for ≥ 1 week before, during, and for ≥ 2 weeks after study completion
* No systemic infection or coagulation disorders
* No psychiatric disturbances that would preclude obtaining informed consent or safe conduct of protocol
* HIV negative
* Hepatitis B surface antigen and hepatitis C antibody negative
* No other active malignancies

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 6 weeks since prior adjuvant radiotherapy or chemoradiotherapy

  * No time restriction for prior curative therapy
* No concurrent pharmacological doses of steroids in any form (topical or systemic)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-09; Primary Completion 2011-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Toxicity profile and overall toxicity rates
Immunologic response rate as measured by ELISPOT assay prevaccination and at days 14 and 18
Biologic response rate

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Ferris, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Cancer Centers, Pittsburgh, Pennsylvania, United States